CLINICAL TRIAL: NCT02377245
Title: Setting up a Pediatric Cohort for Inflammatory Rheumatic Diseases
Brief Title: Juvenile Inflammatory Rheumatism (JIR) Cohorte
Acronym: JIR-cohorte
Status: Enrolling by invitation | Type: Observational
Sponsor: Michaël Hofer (Other)
Collaborators: Hospices Civils de Lyon (Other); Versailles Hospital (Other); Tenon Hospital, Paris (Other); Bicetre Hospital (Other); University of Lausanne Hospitals (Other); University Hospital Muenster (Other); Fondation Rhumatismes-Enfants-Suisse (Unknown)
Responsible Party: Sponsor-Investigator, Michaël Hofer, Head of Pediatric Rheumatology unit, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: JIR-001
Record Dates: First submitted 2014-10-09; First posted 2015-03-03 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Juvenile; Inflammatory; Rheumatism; Pediatric-Onset inflammatory diseases
MeSH Terms: conditions — Arthritis, Juvenile; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Juvenile Inflammatory Rheumatism: Juvenile Inflammatory Rheumatism patients

SUMMARY:
The investigators created a cohort of patients with juvenile inflammatory rheumatisms with the purpose to follow them prospectively, and investigate the tolerance and efficacy of immunosuppresive and biological agents.

DETAILED DESCRIPTION:
The JIR-cohort has to be filled by an authorized investigator during or after the consultation. Each patient much be followed at least once a year.

Different data are requested in the JIR-cohort: diagnosis, treatment, adverse events and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with juvenile inflammatory diseases
* Age at onset up to 18 years old
* Consent according national codes of ethics and current laws

Exclusion Criteria:

* Non-consent from patients and/or legal representative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with juvenile inflammatory diseases
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2014-01; Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of severe and very severe adverse event as a mesure of safety and tolerability | 10 years
Number of treatments prescribed off label | 10 Years
Length in months of drug survival in patient treated with at least two consecutive biological agents | 10 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hofer, Study Director — University of Lausanne Hospitals; Véronique Hentgen, Study Director — Versailles Hospital
Locations (45):
- Belgium (5):
  - Hôpital Reine Fabiola, Brussels
  - CHU Charleroi, Charleroi
  - UZ Leuven, Leuven
  - CHC Liège, Liège
  - CHR Citadelle, Liège
- France (25):
  - CHU Belfort, Belfort
  - CHRU Besançon, Besançon
  - Hôpital Pellegrin enfants, Bordeaux
  - CHRU Brest, Brest
  - Hôpital Femme Mère Enfant, Bron
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Hôpital Nord Marseille, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - Centre hospitalier de Mulhouse, Mulhouse
  - CHU Nantes, Nantes
  - Nice CHU - Lenval, Nice
  - CHU Nimes, Nîmes
  - Hôpital necker Enfants Malade, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Tenon, Paris
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU St-Etienne, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital des enfants, Toulouse
  - CHU Tours, Tours
  - Hôpital André Mignot, Versailles
- University Hospital Muenster, Münster, Germany
- Hôpital Ibnou Rochd, Casablanca, Morocco
- Switzerland (13):
  - CHUV, Lausanne, Canton of Vaud
  - Kantonsspital Aarau, Aarau
  - Kinderspital Basel, Basel
  - Universitäts-Augenklinik Basel, Basel
  - Ospedale Regionale di Bellinzona e valli, Bellinzona
  - Kantonspital Graubunden, Chur
  - Hôpital Ophtalmique, Lausanne
  - Kinderspital Luzern, Lucerne
  - Ospedale Regionale di Lugano, Lugano
  - Ostschweizer Kinderspital St-Gallen, Sankt Gallen
  - Klinik für Rheumatologie und internistische Rehabilitation, Valens
  - Kantonspital Winterthur, Winterthur
  - Kinderspital Zürich, Zurich

REFERENCES:
- [Derived] Pouletty M, Borocco C, Ouldali N, Caseris M, Basmaci R, Lachaume N, Bensaid P, Pichard S, Kouider H, Morelle G, Craiu I, Pondarre C, Deho A, Maroni A, Oualha M, Amoura Z, Haroche J, Chommeloux J, Bajolle F, Beyler C, Bonacorsi S, Carcelain G, Kone-Paut I, Bader-Meunier B, Faye A, Meinzer U, Galeotti C, Melki I. Paediatric multisystem inflammatory syndrome temporally associated with SARS-CoV-2 mimicking Kawasaki disease (Kawa-COVID-19): a multicentre cohort. Ann Rheum Dis. 2020 Aug;79(8):999-1006. doi: 10.1136/annrheumdis-2020-217960. Epub 2020 Jun 11. PMID 32527868
- See also: Official jir-cohorte project webpage — http://www.jircohorte.org